CLINICAL TRIAL: NCT00411528
Title: A Randomized Multicenter Phase II Trial of Patupilone (EPO906) Plus Prednisone Versus Docetaxel Plus Prednisone in Patients With Metastatic Hormone Refractory Prostate Cancer
Brief Title: Efficacy and Safety of Patupilone in Men (≥18 Years) With Metastatic Hormone Refractory Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEPO906A2229; 2006-001822-23 (EudraCT Number)
Record Dates: First submitted 2006-12-12; First posted 2006-12-14 (Estimated); Last update posted 2020-12-17 (Actual); Status verified 2020-09

CONDITIONS: Metastatic Hormone Refractory Prostate Cancer
Keywords: Prostate Cancer; Hormone Refractory; patupilone; docetaxel
MeSH Terms: conditions — Prostatic Neoplasms | interventions — epothilone B; Prednisone; Docetaxel

ARMS (4):
- 1: 8 mg/m2 study drug + prednisone (Experimental): Patupilone 8 mg/m2 + prednisone 5 mg bid daily
  Interventions: Drug: Patupilone; Drug: prednisone
- 2: study drug + prednisone days 1 -8 (Experimental): Patupilone 10 mg/m2 + prednisone days 1 -8 at 25 mg bid, day 9 at 20 mg bid, day 10 at 15 mg bid, day 11 at 10 mg bid, day 12 - 21 at 5 mg bid
  Interventions: Drug: Patupilone; Drug: prednisone
- 3: Study drug + prednisone days 1 - 4 (Experimental): Patupilone 10 mg/m2 + prednisone days 1 - 4 at 5 mg bid, days 5 -12 at 25 mg bid, day 13 at 20 mg bid, day 14 at 15 mg bid, day 15 at 10 mg bid, day 16 - 21 at 5 mg bid
  Interventions: Drug: Patupilone; Drug: prednisone
- 4: Docetaxel 75 mg/m2 + prednisone 5 mg bid daily (Active Comparator): Docetaxel 75 mg/m2 once every 3 weeks + prednisone 5 mg bid daily
  Interventions: Drug: prednisone; Drug: docetaxel

INTERVENTIONS:
Drug: Patupilone
  Other Names: EPO906
  Arms: 1: 8 mg/m2 study drug + prednisone; 2: study drug + prednisone days 1 -8; 3: Study drug + prednisone days 1 - 4
Drug: prednisone
Drug: docetaxel
  Arms: 4: Docetaxel 75 mg/m2 + prednisone 5 mg bid daily

SUMMARY:
The objective of this study is to assess the response of patupilone plus prednisone compared to docetaxel plus prednisone on prostate specific antigen (PSA) in patients with metastatic hormone refractory prostate cancer. Additionally, this study will assess the response on measureable disease and the effects on patient-reported outcomes.

ELIGIBILITY:
Inclusion criteria:

* Must be ≥ 18 years of age
* Confirmed and documented diagnosis of prostate cancer
* Confirmed and documented evidence of progression of disease (hormone refractory)
* Low testosterone levels
* Chemotherapy-naïve

Exclusion criteria:

* Recent radiation therapy (within 4 weeks)
* Known brain metastasis
* Peripheral neuropathy
* Active diarrhea
* Significant illnesses such as heart disease, diabetes, or chronic or uncontrolled infections
* Allergic reactions to patupilone or docetaxel or prednisone or similar compounds

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2006-09; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Antitumor response based on PSA decrease | Every 3 weeks

SECONDARY OUTCOMES:
Measurable soft tissue response for both regimens | Every 6 weeks or every 12 weeks if patient has bone disease for bone scan

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (30):
- United States (11):
  - University of California San Diego Dept of Moores Cancer Center, La Jolla, California
  - University of Colorado Dept. of Univ. of Colorado, Aurora, Colorado
  - Norwalk Hospital, Norwalk, Connecticut
  - Georgetown University/Lombardi Cancer Center Dept.of Lombardi Cancer Center, Washington D.C., District of Columbia
  - MD Anderson Cancer Center - Orlando CEPO906A2229, Orlando, Florida
  - H. Lee Moffitt Cancer Center/University of South Florida Department of Genitourology, Tampa, Florida
  - Palm Beach Cancer Institute, West Palm Beach, Florida
  - NorthWest Georgia Oncology Centers Marietta Center, Marietta, Georgia
  - University Chicago Hospital StudyCoordinator:CEPO906A2229, Chicago, Illinois
  - Queens Cancer Center of Queens Hospital, Jamaica, New York
  - Oregon Health & Science University StudyCoordinator:CEPO906A2229, Portland, Oregon
- Australia (3):
  - Novartis Investigative Site, Kogarah, New South Wales
  - Novartis Investigative Site, South Brisbane, Queensland
  - Novartis Investigative Site, Parkville, Victoria
- Novartis Investigative Site, Ghent, Belgium
- France (6):
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Colmar
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Rouen
  - Novartis Investigative Site, Strasbourg
  - Novartis Investigative Site, Toulouse
- Germany (2):
  - Novartis Investigative Site, Mannheim
  - Novartis Investigative Site, Weiden
- Italy (2):
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Perugia, PG
- Novartis Investigative Site, Singapore, Singapore
- Spain (4):
  - Novartis Investigative Site, Málaga, Andalusia
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, Madrid

REFERENCES:
- [Derived] de Liano AG, Reig O, Mellado B, Martin C, Rull EU, Maroto JP. Prognostic and predictive value of plasma testosterone levels in patients receiving first-line chemotherapy for metastatic castrate-resistant prostate cancer. Br J Cancer. 2014 Apr 29;110(9):2201-8. doi: 10.1038/bjc.2014.189. Epub 2014 Apr 10. PMID 24722180
- See also: Visit NovartisClinicalTrials.com: Pre-qualify for a trial, and view a list of trials and participating study centers. — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=8483